CLINICAL TRIAL: NCT06994052
Title: A Phase Ⅳ Clinical Trial to Evaluate the Immunogenicity and Safety of Booster Immunization With Varicella Vaccine at Different Intervals Among Children Aged 7-12 Years
Brief Title: Study on Booster Immunization With Varicella Vaccine at Different Intervals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-VAR-MA4004-JS-1
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: VZV; Varicella Immunisation
MeSH Terms: interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Participants received a single dose of varicella vaccine as booster immunization 3 months after their primary vaccination.
  Interventions: Biological: Varicella vaccine
- Group B (Experimental): Participants received a single dose of varicella vaccine as booster immunization 18-30 months after their primary vaccination.
  Interventions: Biological: Varicella vaccine
- Group C (Experimental): Participants received a single dose of varicella vaccine as booster immunization 36-48 months after their primary vaccination.
  Interventions: Biological: Varicella vaccine
- Group D (Experimental): Participants received a single dose of varicella vaccine as booster immunization 60-72 months after their primary vaccination.
  Interventions: Biological: Varicella vaccine

INTERVENTIONS:
Biological: Varicella vaccine — lyophilized powder, subcutaneous injection

SUMMARY:
The goal of this clinical trial is to evaluate the immunogenicity and safety of booster immunization of varicella live attenuated vaccine (varicella vaccine hereafter) at different intervals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 7-12 years;
* Has previously received a single dose of varicella vaccine, with at least 3 months since the first dose;
* The subject or legal guardian can understand and sign the informed consent form (double signature is required for those over 8 years old);
* Participants and their legal guardians voluntarily participate in the study and are able to comply with all study procedures;
* Provide legal identity proof;

Exclusion Criteria:

* History of varicella;
* History of severe allergic reactions to vaccines (such as acute anaphylaxis, angioedema, dyspnea, etc.);
* Suffering from acute disease, severe chronic disease, acute exacerbation of chronic disease;
* With any confirmed or suspected immunodeficiency disease, immunocompromised or receiving immunosuppressive therapy (including systemic steroid therapy);
* With a history of congenital immune diseases or close contact with family members with a history of congenital immune diseases;
* With encephalopathy, uncontrolled epilepsy, other progressive neurological disorders, history of Guillain-Barre syndrome;
* Body temperature >37℃ at the time of vaccination;
* Receipt of blood products within 3 months before receiving investigational vaccine;
* Receipt of another study drug within 30 days before receipt of the investigational vaccine;
* Receipt of live attenuated vaccine within 28 days before receipt of investigational vaccine;
* Receipt of subunit or inactivated vaccine within 7 days before receipt of investigational vaccine;
* Participated in other clinical trials before enrollment and were enrolled in another clinical trial during the follow-up period or planned to participate in another clinical trial within 3 months;
* The participant had any other factors that were ineligible for vaccination by in the investigator's judgment.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 412 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of varicella-zoster virus (VZV) antibodies | 30 days after booster dose immunization
  GMT of VZV antibodies 30 days after booster dose immunization

SECONDARY OUTCOMES:
Seroconversion rate of varicella-zoster virus (VZV) antibodies | 30 days after booster dose immunization
  Seroconversion rate of VZV antibodies 30 days after booster dose immunization
Seropositive rate of varicella-zoster virus (VZV) antibodies | 30 days after booster dose immunization
  Seropositive rate of VZV antibodies 30 days after booster dose immunization
Geometric mean increase (GMI) of varicella-zoster virus (VZV) antibodies | 30 days after booster dose immunization
  GMI of VZV antibodies 30 days after booster dose immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Disease control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No